CLINICAL TRIAL: NCT00735670
Title: Treatment of Mild to Moderate Depression Symptoms in Patients With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Denise Tate, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NDNO60032SS; NIDRRH133N060032
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Spinal Cord Injury
Keywords: SCI
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Venlafaxine (Experimental): Venlafaxine HCl is classified as a selective serotonin and norepinephrine reuptake inhibitor (SSNRI) and has been approved by the FDA for the treatment of major depressive disorder. The treatment group will receive a sub-therapeutic dose over a two week period, with a two week titration, starting at 37.5 mg up to a maximum dose of 150 mg per day. At the end of the treatment period, dosage was tapered down in a step-wise fashion over a period of three weeks; 75 mg. for two weeks and 37.5 mg. for one week. While this was the standard protocol, study drug tapering was individualized based on side effects and the clinical judgment of the prescriber.
  Interventions: Drug: Venlafaxine HCl
- Placebo (Placebo Comparator): Placebo capsules were compounded by filling a matching gelatin capsule with lactose. Titration up and down followed the same schedule as the treatment group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Venlafaxine HCl — Starting dose is 37.5 mg and ending dose is 150 mg at 13 weeks. From weeks 13 to 26 subjects no longer will receive the drug
  Other Names: Effexor XR
  Arms: Venlafaxine
Other: Placebo — Subjects received a placebo instead of Venlafaxine HCl until week 13 as did the Venlafaxine group.
  Arms: Placebo

SUMMARY:
This study was initially designed to test the efficacy of Venlafaxine HCl in reducing incidence of the onset of major depression after a new spinal cord injury (SCI). After several protocol modifications, the purpose of the study is to test the effectiveness of a sub-therapeutic dose of Venlafaxine HCl to reduce mild to moderate symptoms in persons with SCI.

DETAILED DESCRIPTION:
The successes of psychological and pharmacological modes of intervention in treating depression, both alone and combined, are well documented in the literature. While a great deal of research has identified specific clinical indications for many antidepressants currently available in the general population, little is known about the clinical indications of these agents in SCI. This study is proposed to test the benefits of Venlafaxine HCI (Effexor XR) for reducing mild to moderate symptoms of depression among people with SCI. The intervention will last 12 weeks and there will be 13 assessments and data collection points. Data will be collected at 26 weeks also. Eight face to face contacts are anticipated.

Because of the change in protocol to reducing mild to moderate symptoms and substantially lower enrollment than anticipated (1/6th of what we anticipated), we deleted a number of study outcomes listed in the 2011 posting of this study. Most of these were not part of the original posting in 2008, and those that were deleted were no longer relevant to new protocol's focus on reducing mild to moderate depression. The two outcomes reported here were most relevant to the revised protocol.

ELIGIBILITY:
Inclusion Criteria:

* Having sustained an SCI at least six months prior to enrollment.
* Neurological impairment ASIA Grades A-D.
* Mild to moderate depressive symptoms.
* English speaker
* Age 18 years or older
* Able to communicate with study personnel

Exclusion Criteria:

* No neurological impairment due to SCI.
* Presence of cognitive deficits precluding and giving informed consent and completion of survey based assessment tools.
* Psychiatric contraindications (suicidal ideation, history of suicidal attempts, alcohol and drug dependency, other psychiatric diagnosis including bipolar disorder).
* Medical contraindications (terminal illness or unstable medical condition as determined by medical history and/or examination).
* Pregnant or unwilling to use birth control if female and sexually active.
* Presence of glaucoma.
* Prior use of study drug without success or being treated with another antidepressant medication and being unwilling to taper off to take the stud drug.
* Willing to travel to Ann Arbor Michigan.
* Expecting to take or currently taking another experimental study within 30 days
* Major surgery scheduled within 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-06; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise G Tate, Ph.D., Principal Investigator — University of Michigan Department of Physical Medicine and Rehabilitation; Anthony Chiodo, M.D., Study Director — University of Michigan
Locations (1):
- University of Michigan Model SCI Care System, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment into the final protocol began in May 2009 and continued through July 2011. Participants were recruited from the surrounding community through clinics, existing research studies, and community organizations.
Pre-assignment Details: Because of challenges of recruiting inpatients with new injuries, the final modification to the protocol was to restrict inclusion criteria to those with chronic SCI (>6 months after injury) and the objective of the study shifted from preventing a major depressive episode to a reduction in symptoms. Therefore 13 / 34 enrolled were ineligible.
Period: Overall Study
Arm/Group | Venlafaxine | Placebo
Started | 10 | 11
Completed | 6 | 6
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Population: Participants meeting eligibility criteria for the final protocol version.
Groups:
- Total: Total of all reporting groups
Arm/Group | Venlafaxine | Placebo | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (10.5) | 51.7 (14.1) | 48.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21
Time since injury [Mean (Standard Deviation); unit: years] | 10.01 (9.0) | 13.64 (15.1) | 11.9 (10.0)
Level of injury [Number; unit: participants]
  Tetraplegia | 6 | 1 | 7
  Paraplegia | 4 | 10 | 14

OUTCOME MEASURES:

1. Primary Outcome: 16-Item Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR16)
Description: The QIDS assesses symptoms of depression across the nine DSM-IV criterion domains for major depressive episode. The primary end-point in this study was the number of participants who had a >50% change in scores on the QIDs from baseline to week 13 (end of treatment period).
Time Frame: Baseline and Week 13
Population: Participants who completed the week 13 assessment.
Measure: Number; unit: participants
Arm/Group | Venlafaxine | Placebo
Number analyzed (Participants) | 6 | 6
participants | 2 | 0
Statistical Analysis 1: Comparison: Venlafaxine vs Placebo; Test type: Superiority or Other; p = 0.445, Fisher Exact

2. Secondary Outcome: Depression Scale of the Patient Health Questionnaire (PHQ-9)
Description: The nine items of the PHQ-9 are based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV. Higher total scores indicate more severe symptomatology, ranging from 0 (no symptoms) to 27 (most severe symptoms). Data in the tables begin with the overall mean for each group that includes all subjects, average across all assessment time points. Each subsequent row reports the mean and standard deviation of each time point by allocation, noting sample size for each group in the arm/group title given missing data in each time point after baseline.
Time Frame: Baseline and weeks 1, 2, 3, 5, 9, 13, 14, 15, 16, 18, 20 and 26 weeks
Population: Subjects with PHQ-9 data at any of the measurement time points (baseline, weeks 1, 2, 3, 5, 9, 13, 14, 15, 16, 18, 20 and 26 weeks) are included in the means reported for each time point. The sample size for each time point is given in the category title (e.g., 10Ven = 10 venlafaxine group or 11Plac = 11 placebo group) if it deviates from baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venlafaxine | Placebo
Number analyzed (Participants) | 10 | 11
units on a scale
  Overall Mean | 4.84 (3.66) | 5.46 (4.48)
  Baseline | 8.9 (1.12) | 10.36 (3.58)
  Week 1 (7Ven, 6Plac) | 7 (3.36) | 9.67 (2.94)
  Week 2 (6Ven, 6Plac) | 4.5 (2.16) | 5.00 (4.14)
  Week 3 (6Ven, 6Plac) | 2.67 (1.96) | 5.00 (4.00)
  Week 5 (6Ven, 6Plac) | 4.33 (2.58) | 3.83 (3.37)
  Week 9 (5Ven, 7Plac) | 4.80 (2.68) | 4.71 (5.12)
  Week 13 (6Ven, 6Plac) | 5.67 (5.1) | 3.33 (4.36)
  Week 14 (4Ven, 6Plac) | 4.25 (2.21) | 4.17 (4.31)
  Week 15 (5Ven, 5 Plac) | 1.80 (1.30) | 3.20 (3.96)
  Week 16 (4Ven, 6 Plac) | 2.00 (1.41) | 3.20 (4.14)
  Week 18 (4Ven, 5Plac) | 2.25 (2.21) | 4.00 (3.08)
  Week 20 (6Ven, 4Plac) | 3.67 (3.98) | 4.75 (4.64)
  Week 26 (6Ven, 5Plac) | 5.50 (3.67) | 4.40 (4.27)
Statistical Analysis 1: Comparison: Venlafaxine vs Placebo; A linear mixed model (LMM) analysis was used and included a random intercept effect based on lowest Akaike's Information Criterion values when we compared three random coefficient models (intercept, slope and intercept and slope). To examine whether allocation group influenced the effect of time and baseline PHQ-9 sore on the trajectory of PHQ-9 scores, we included two interaction terms (time by allocation group and baseline PHQ-9 score by allocation group); Test type: Superiority or Other; p = 0.725, Mixed Models Analysis — Comparison of venlafaxine vs. placebo on change of PHQ-9 over time controlling for baseline PHQ-9 score; REML = -0.31, 95% CI 2-sided [-0.48 to -0.15]

ADVERSE EVENTS:
Time Frame: May 2009 through January 2012
Arm/Group | Venlafaxine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/11
Other Adverse Events (participants affected / at risk) | 4/10 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venlafaxine (N=10) | Placebo (N=11)
kidney infection (unrelated) (Renal and urinary disorders) | 1 (1) | 0 (0) — Subject was hospitalized with kidney infection which was determined to be unrelated to the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venlafaxine (N=10) | Placebo (N=11)
Side effects (General disorders) | 3 (3) | 4 (4) — Includes side effects of feeling "spacey", sleepiness, drowsiness, sexual dysfunction, irritability.
Onset of major depressive episode (Psychiatric disorders) | 0 (0) | 1 (1)
Suddenly stopped taking medication (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Difficulties with recruitment and high rate of withdrawal (57%) resulted in a very small sample. As such, results must be taken with caution given low power in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes